CLINICAL TRIAL: NCT05643560
Title: Long-term Treatment Outcome of Jivi® Prophylaxis on Joint Health in Adult Patients With Hemophilia A
Brief Title: An Observational Study Called JOIHA to Learn More About How Well the Treatment With Jivi Works to Prevent Problems With Joints in Adults With Hemophilia A.
Acronym: JOIHA
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22082
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A; Prophylaxis of Bleeding
Keywords: Joint health; Hemophilia A; Clotting factor VIII (FVIII); Physical activity
MeSH Terms: conditions — Hemophilia A; Motor Activity | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients: Hemophilia patients who had initiated damoctocog alfa pegol treatment .
  Interventions: Drug: Damoctocog alfa pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, BAY94-9027) — Intervention is given as part of routine medical practice.

SUMMARY:
This is an observational study in which data from people with hemophilia A who decide on their own or by recommendation of their doctors to take Jivi are collected and studied. In observational studies, only observations are made without specified advice or interventions.

Hemophilia A is a genetic bleeding disorder that is caused by the lack of a protein in the blood called "clotting factor 8" (FVIII). FVIII is naturally found in the blood where it causes the blood to clump together to help prevent and stop bleeding. People with lower levels of FVIII or with FVIII that does not work properly may bleed for a long time from minor wounds, have painful bleeding into joints, or have internal bleeding.

The study treatment, Jivi (also called damoctocog alfa pegol), is already available for doctors to prescribe to people with hemophilia A to treat and prevent bleeding. It works by replacing the missing FVIII, or the FVIII that does not work properly.

People with hemophilia A need frequent injections of FVIII products into the vein. So called standard half-life (SHL) products need to be given 2 to 4 times a week for the prevention of bleeding. In recent years, new products like Jivi called extended half-life (EHL) products have available. These products last longer in the body so that they require to be given less often with injections up to every 7 days. Thus, these treatments may be easier and more comfortable to stick to in daily life. There is no general plan concerning the best amount of treatment and the frequency of injections for the prevention of bleeding, since the severity may be different and individual risk factors have to be considered. Doctors often decide on a treatment plan based on patient's disease and response.

Clinical studies have already shown that people with hemophilia A benefit from the treatment with Jivi. However, there are no data available coming from the real-world about how well Jivi works to support joint health, measured by ultrasound (US) examination and HEAD-US score.

In this study, researchers want to learn more about how well Jivi works if used for prolonged periods of treatment under real-world settings to prevent problems with joints in people with hemophilia A. How well it works means to find out if participants' joints status can be improved by treatment with Jivi.

To do this, researchers will collect data about participants' joints status by

* making images of participants' joints by using sound waves (ultrasound), and
* using HEAD-US score after 24 months of treatment with Jivi. The researchers will then compare these data to the participants' joints status before treatment start with Jivi.

Besides this data collection, no further tests or examinations are planned in this study.

Some participants in this study will already be receiving treatment with Jivi as part of their regular care no more than 12 months. And some participants will start to take Jivi in this study as prescribed by their doctors during routine practice according to the approved product information.

The researchers will collect data from each patient for a period of 26 months after initiation of the Jivi treatment.

There are no required visits or tests in this study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis hemophilia A with FVIII:C ≤2%.
* Patients ≥ 18 years of age.
* Previously treated for hemophilia A (PTPs).
* Patients who had initiated damoctocog alfa pegol maximum 12 months prior to enrollment into the study or who initiate damoctocog alfa pegol treatment at the enrollment , where the decision to initiate damoctocog alfa pegol has been made before the decision for study participation.
* Patients having a HEAD-US measurement available in the 2 months prior to damoctocog alfa pegol treatment initiation.
* Patients without previous history of FVIII inhibitors or patients with previous history of FVIII inhibitors on standard prophylaxis therapy for at least 1 year prior to baseline (damoctocog alfa pegol treatment initiation).
* No current evidence of FVIII inhibitor or clinical suspicion of FVIII inhibitor.
* Signed informed consent/assent.

Exclusion Criteria:

* Concurrent participation in an investigational program with interventions outside of routine clinical practice.
* Diagnosis of any other bleeding/coagulation disorder other than hemophilia A.
* Patient on immune tolerance induction (ITI) treatment at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who initiate damoctocog alfa pegol treatment at the enrollment or who had initiated damoctocog alfa pegol treatment maximum 12 months prior to enrollment and having a HEAD-US score measurement available within 2 months prior to damoctocog alfa pegol initiation.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an unchanged or decreased HEAD-US score at 24 months after treatment initiation with damoctocog alfa pegol | 24 months
  The Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) score is based on the three markers for the main joints (knees, elbows, ankles): synovitis (score: 0-2), cartilage (score: 0-4), subchondral bone (score: 0-2).

SECONDARY OUTCOMES:
Occurrence of an unchanged or decreased HEAD-US score at 12 months after treatment initiation with damoctocog alfa pegol | 12 months
Occurrence of a decrease in joint ABR together with a decrease in HEAD-US score 12 and 24 months after treatment initiation with damoctocog alfa pegol | 12 months and 24 months
  ABR: Annualized bleeding rate.
Change in the number of target joints (as defined by ISTH) 12 months and 24 months after treatment initiation with damoctcog alfa pegol in relation to HEAD-US score | From baseline to 12 months and 24 months
  ISTH: International Society on Thrombosis and Hemostasis.
Change in HEAD-US score and HJHS score 12 months and 24 months after treatment initiation with damoctocog alfa pegol | From baseline to 12 months and 24 months
  The Hemophilia Joint Health Score (HJHS) measures joint health, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia: the knees, ankles, and elbows.
Change in physical activity (IPAQ-SF) 12 months and 24 months after treatment initiation with damoctocog alfa pegol by categorized HEAD-US score change | From baseline to 12 months and 24 months
  The International Physical Activity and sports short form (IPAQ-SF) questionnaire consists of 7 items and will ask about the time one spent being physically active in the last 7 days.
Change in pain (Visual Analogue Scale) 12 months and 24 months after treatment initiation with damoctocog alfa pegol by categorized HEAD-US score change | From baseline to 12 months and 24 months
  Pain Visual Analogue Scale (VAS) score categorized as "no pain (0-4)", "mild pain (5-44)", "moderate pain (45-74)" and "severe pain (75-100)" vs. HEAD-US score change categories (worsened, unchanged, improved).

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Italy

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.